CLINICAL TRIAL: NCT04680221
Title: Stopping Opioid Overuse in Obstetrics to Halt Exposure Trial
Acronym: SOOOTHE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Collaborators: Truman Medical Center (Other)
Responsible Party: Principal Investigator, Traci N Johnson, Principal Investigator, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2026221; 21-018 (Other: Truman Medical Center)
Record Dates: First submitted 2020-10-29; First posted 2020-12-22 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Pain, Postoperative; Opioid Use
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment (Active Comparator): The transversus abdominis plane block is a procedure involving injection of a local anesthetic solution into the abdominal plane between the internal oblique muscle and the transversus abdominis muscle. In our institution, this is done under ultrasound guidance which is the current standard to improve efficacy and limit complications. Liposomal bupivacaine uses an innovative technology consisting of lipid-based particles containing active pharmaceutical agent (bupivacaine) which extends the duration of the medication through a process of gradual release for metabolism.This drug delivery technology extends the duration of action to up to 96 hours when given at a dose of 266 mg liposomal bupivacaine admixed with 30 ml of bupivacaine 0.25% and 30 ml of saline. Forty ml of solution is deposited on the left side of the abdomen and 40 ml on the right.
  Interventions: Drug: Liposomal bupivacaine; Procedure: TAP block
- Control (Placebo Comparator): The transversus abdominis plane block will be performed under ultrasound guidance with deposition of 80 ml of saline (40 ml on either side).
  Interventions: Procedure: TAP block; Drug: Deposition of saline

INTERVENTIONS:
Drug: Liposomal bupivacaine — Deposition of liposomal bupivacaine
  Other Names: EXPAREL
  Arms: Treatment
Procedure: TAP block — Transversus abdominis plane block performed to deposit anesthetic
Drug: Deposition of saline — Deposition of saline
  Arms: Control

SUMMARY:
As the opioid epidemic continues on, more research is needed on multi-modal approaches to decrease opioid exposure after common procedures. The aim of this study is to investigate the role of a transverses abdominis block using liposome bupivacaine suspension in reducing use of opioid medications through post-operative day 7. The study is a proposed double-blind, randomized controlled trial.

DETAILED DESCRIPTION:
Nearly 1 in 3 women in the US deliver by cesarean delivery. After cesarean delivery, approximately 75-87% percent of women are discharged from the hospital with an opioid prescription. Most women fill that prescription and 1% continue to use those opioids 90 days after delivery despite no longer requiring them for pain control, predisposing them to opioid dependence. This study aims to determine if transverse abdominis plane (TAP) block using bupivacaine liposome suspension injection (EXPAREL®) significantly reduces the use of opioid medications after discharge in women undergoing scheduled cesarean delivery. The study is a proposed double-blinded, randomized controlled trial. Pregnant women who have completed 37 weeks gestation and are scheduled for cesarean delivery will be randomized to receive a TAP block with 80 ml of mixed liposomal bupivacaine or saline. Based on its use in other surgical settings, the investigators hypothesize that women who receive a liposomal bupivacaine TAP block will use significantly less opioids by postoperative day 7 as calculated in morphine milligram equivalents. In addition to overall consumption of opioids after discharge, other aims to be studied include inpatient opioid use, effect on pain scores, rates of postpartum depression, patient-perceived quality of breastfeeding, patient quality of recovery, and composite adverse outcomes.

With better overall pain control and less dependence on opioids postpartum, liposomal bupivacaine TAP blocks at the time of scheduled cesarean delivery may offer a highly effective analgesic alternative that can help shift the tide in the ongoing opioid epidemic among reproductive females.

ELIGIBILITY:
Inclusion Criteria:

* Unlabored, scheduled primary or repeat cesarean delivery
* Cesarean performed by obstetrician or surgically-trained family medicine physician
* Ability to complete numeric pain scale assessment and surveys
* Patients who do not speak English but are able to converse via an interpreter both in person and by phone

Exclusion Criteria:

* Complications requiring return to the operating room
* Unscheduled deliveries
* <18 years old, >45 years old
* Twin deliveries
* Preterm deliveries (<37 wks)
* Current or previous history of opioid-substance use disorder according to patient report or medical chart
* Prescription of opioid medication filled in previous 30 days prior to delivery according to patient report, documentation in electronic medical record, or documentation in the prescription drug monitoring program
* Allergy to local anesthetics or NSAIDs
* Cardiovascular disease, eg arrhythmia, or ASA (American Society of Anesthesiologists) Class III or higher
* Diagnosis of liver disorder or dysfunction including fatty liver of pregnancy, preeclampsia with severe features including liver or kidney involvement
* Known significant renal disease, oliguria, or Cr >1.1.
* Platelet count less than or equal to 90k or rapid decline in third trimester or other coagulopathy
* Infection overlying the regional anesthesia site
* Hypovolemia prohibiting regional anesthesia
* General anesthesia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Morphine Milligram Equivalents | 7 days after cesarean
  Amount of opioid medications taken converted to Morphine Milligram Equivalents

SECONDARY OUTCOMES:
Morphine Milligram Equivalents at 48 hours | Time surgery is complete to 48 hours
  Total opioid use inpatient at 48 hours as measured in Morphine Milligram Equivalents
Numeric Rating Scale Pain Score on postoperative day 1 | Midnight to midnight postoperative day #1
  Highest documented pain score postoperative day #1 by Numeric Rating Scale Pain level [0-10]. Higher scores denote more pain.
Time to as needed opioid use | Inpatient stay up to 6 days
  Time to first "as needed" opioid use while inpatient
Opioid-spared Percentage | Inpatient stay up to 6 days
  Percentage of patients in each arm that did not receive any additional opioid after surgery
Edinburgh Postpartum Depression Scale Score at Discharge | Inpatient stay up to 6 days
  Score on the Edinburgh Postpartum Depression scale [0-30] at discharge. Higher scores denote worse depression. A positive question 10 is also positive.
Edinburgh Postpartum Depression Scale Score at 7 days | Postoperative day #7
  Score on the Edinburgh Postpartum Depression scale [0-30] by phone interview postoperative day #7. Higher scores denote worse depression. A positive question 10 is also positive.
Edinburgh Postpartum Depression Scale Score at 14 days | Postoperative day #14
  Score on the Edinburgh Postpartum Depression scale [0-30] at appointment postoperative day #14. Higher scores denote worse depression. A positive question 10 is also positive.
Edinburgh Postpartum Depression Scale Score at 6 wks | 6 weeks postpartum visit
  Score on the Edinburgh Postpartum Depression scale [0-30] at 6 week postoperative appointment. Higher scores denote worse depression. A positive question 10 is also positive.
Numeric Rating Scale Pain Score Postoperative day #7 | Postoperative day #7
  Numeric Rating Scale Pain level [0-10] assessed by phone interview on Postoperative day #7. Higher scores denote more pain.
Numeric Rating Scale Pain Score at Postoperative day #14 | Postoperative day #14
  Numeric Rating Scale Pain level [0-10] at 2 week post op visit. Higher scores denote more pain.
Numeric Rating Scale Pain Score at 6 wks | Postpartum visit 6 wks
  Numeric Rating Scale Pain level [0-10] at 6 week post op visit. Higher scores denote more pain.
Quality of Recovery-15 at discharge | Inpatient stay up to 6 days
  Quality of Recovery scale at discharge
Quality of Recovery-15 at 7 day | Postoperative day #7
  Quality of Recovery scale at Postoperative day #7 by phone interview [0-150].The Quality of Recovery-15 scores for excellent, good, moderate, and poor recovery were 136-150, 122-135, 90-121, and 0-89, respectively.
Quality of Recovery-15 at Postoperative day #14 | Postoperative day #14
  Quality of Recovery scale at post op visit [0-150]. The Quality of Recovery-15 scores for excellent, good, moderate, and poor recovery were 136-150, 122-135, 90-121, and 0-89, respectively.
Quality of Recovery-15 at 6 weeks | Postpartum visit 6 weeks
  Quality of Recovery scale at postpartum visit [0-150].The Quality of Recovery-15 scores for excellent, good, moderate, and poor recovery were 136-150, 122-135, 90-121, and 0-89, respectively.
Breastfeeding Self-Efficacy Scale Short Form at Postoperative day #7 | Postoperative day #7
  Breastfeeding Self-Efficacy Scale Short Form at Postoperative day #7 by phone interview [14-70] with higher scores denoting higher confidence
Breastfeeding Self-Efficacy Scale Short Form at Postoperative day #14 | Postoperative day #14
  Breastfeeding Self-Efficacy Scale Short Form at post op visit [14-70] with higher scores denoting higher confidence
Breastfeeding Self-Efficacy Scale Short Form at 6 weeks | Postpartum 6 weeks
  Breastfeeding Self-Efficacy Scale Short Form at postpartum visit [14-70] with higher scores denoting higher confidence
Adverse Events | Study duration ~ 8 weeks
  Adverse outcomes or side effects

CONTACTS AND LOCATIONS:
Overall Officials: Devika Maulik, MD, Study Chair — Children's Mercy Hospital Kansas City; Gary Sutkin, MD, Study Chair — University of Missouri, Kansas City
Locations (1):
- Truman Medical Center - Lakewood, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin JA, Hamilton BE, Osterman MJK, Driscoll AK. Births: Final Data for 2018. Natl Vital Stat Rep. 2019 Nov;68(13):1-47. PMID 32501202
- [Background] Peahl AF, Dalton VK, Montgomery JR, Lai YL, Hu HM, Waljee JF. Rates of New Persistent Opioid Use After Vaginal or Cesarean Birth Among US Women. JAMA Netw Open. 2019 Jul 3;2(7):e197863. doi: 10.1001/jamanetworkopen.2019.7863. PMID 31348508
- [Background] Badreldin N, Grobman WA, Chang KT, Yee LM. Opioid prescribing patterns among postpartum women. Am J Obstet Gynecol. 2018 Jul;219(1):103.e1-103.e8. doi: 10.1016/j.ajog.2018.04.003. Epub 2018 Apr 7. PMID 29630887
- [Background] Bateman BT, Franklin JM, Bykov K, Avorn J, Shrank WH, Brennan TA, Landon JE, Rathmell JP, Huybrechts KF, Fischer MA, Choudhry NK. Persistent opioid use following cesarean delivery: patterns and predictors among opioid-naive women. Am J Obstet Gynecol. 2016 Sep;215(3):353.e1-353.e18. doi: 10.1016/j.ajog.2016.03.016. Epub 2016 Mar 17. PMID 26996986
- [Background] Tuthill EL, McGrath JM, Graber M, Cusson RM, Young SL. Breastfeeding Self-efficacy: A Critical Review of Available Instruments. J Hum Lact. 2016 Feb;32(1):35-45. doi: 10.1177/0890334415599533. Epub 2015 Aug 28. PMID 26319113
- [Background] Dennis CL. The breastfeeding self-efficacy scale: psychometric assessment of the short form. J Obstet Gynecol Neonatal Nurs. 2003 Nov-Dec;32(6):734-44. doi: 10.1177/0884217503258459. PMID 14649593
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Background] Eisenach JC, Pan PH, Smiley R, Lavand'homme P, Landau R, Houle TT. Severity of acute pain after childbirth, but not type of delivery, predicts persistent pain and postpartum depression. Pain. 2008 Nov 15;140(1):87-94. doi: 10.1016/j.pain.2008.07.011. Epub 2008 Sep 24. PMID 18818022
- [Background] Babazade R, Vadhera RB, Krishnamurthy P, Varma A, Doulatram G, Saade GR, Turan A. Acute postcesarean pain is associated with in-hospital exclusive breastfeeding, length of stay and post-partum depression. J Clin Anesth. 2020 Jun;62:109697. doi: 10.1016/j.jclinane.2019.109697. Epub 2019 Dec 31. PMID 31899076
- [Background] Mustafa HJ, Wong HL, Al-Kofahi M, Schaefer M, Karanam A, Todd MM. Bupivacaine Pharmacokinetics and Breast Milk Excretion of Liposomal Bupivacaine Administered After Cesarean Birth. Obstet Gynecol. 2020 Jul;136(1):70-76. doi: 10.1097/AOG.0000000000003886. PMID 32541292
- [Background] Hebbard P, Fujiwara Y, Shibata Y, Royse C. Ultrasound-guided transversus abdominis plane (TAP) block. Anaesth Intensive Care. 2007 Aug;35(4):616-7. No abstract available. PMID 18020088
- See also: CDC Guideline for Prescribing Opioids for Chronic Pain - United States, 2016 — https://www.cdc.gov/mmwr/volumes/65/rr/rr6501e1.htm